CLINICAL TRIAL: NCT03304119
Title: Torsion of the Tibial Tuberosity, a New Factor of Patellar Instability?
Status: Completed | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Vincent Chassaing (Unknown); European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: RGDS TTA study
Record Dates: First submitted 2017-09-26; First posted 2017-10-06 (Actual); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2018-02

CONDITIONS: Patellar Instability; Patellar Dislocation
Keywords: Torsion of tibial tuberosity; Recurrent patellar dislocation; MRI Measurements; Patellar instability; Patellar dislocation; Tibial tubercle position; Tibial tubercle torsion
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patellar instability group: Group of patients with patellar instability stemming from a recurrent patellar dislocation
- Control group control: Group that has not been checked for patellar instability.

SUMMARY:
Patellar instability (recurrent patellar dislocation) can occur at any age. It is most often seen in young subjects, especially among adolescents. It is commonly accompanied by anatomical factors. A new factor not described in bibliographic sources and characterized by an external torsion of the tibial tuberosity is frequently found in patients with patellar instability thanks to MRIs. This does not seem to be the case when there is no patellar pathology. A statistical study is needed to assess this rotary anomaly. Validate the predictive benefits when measuring the torsion of tibial tuberosity in cases with recurrent patellar dislocation.

DETAILED DESCRIPTION:
Patellar instability (recurrent patellar dislocation) can occur at any age. It is most often seen in young subjects, especially among adolescents. It is commonly accompanied by anatomical factors known to be driving: Dysplasia of the trochlea, patella alta, lateralisation of the tibial tuberosity, patellar torsion and misalignment, tearing of the Medial Patello Femoral Ligament... The assessment of these factors is essential to evaluate the instability and guide the procedures of the surgical treatment. MRIs have become an important test for the analysis and measurement of these factors. A new factor not described in bibliographic sources and characterized by an external torsion of the tibial tuberosity is frequently found in patients with patellar instability thanks to MRIs. This does not seem to be the case when there is no patellar pathology. A statistical study is needed to assess this rotary anomaly. It will be necessary to take it into account in the future regarding indications and techniques for tibial tuberosity osteotomies, often used to correct patellar instability.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Subjects who have not expressed opposition to the use of the data for research purposes

Clinical criteria:

* Unstable group:

  * Medical history with 2 patellar dislocations or more,
  * with or without requiring surgical treatment after an MRI Control group: Men or women over 18 years old
  * Subjects who have not expressed opposition to the use of the data for research purposes
* Control group:

  * Patients showing meniscal injury on MRI who may or may not have been treated (meniscectomy or stitches)

Exclusion Criteria:

* Unstable group:

  * MRI performed on one knee operated for patellar instability
  * Associated tearing of the ligament (ACL, PCL)
* Control group:

  * Patients with a medical history of patellar pathology
  * Patients with associated ligament injury (ACL, PCL)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: group of patients with patellar instability stemming from a recurrent patellar dislocationand a control group that has not been checked for patellar instability.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ECTEN, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skelley N, Friedman M, McGinnis M, Smith C, Hillen T, Matava M. Inter- and intraobserver reliability in the MRI measurement of the tibial tubercle-trochlear groove distance and trochlea dysplasia. Am J Sports Med. 2015 Apr;43(4):873-8. doi: 10.1177/0363546514565768. Epub 2015 Jan 28. PMID 25632054
- [Background] The Patellofemoral Joint - State of the Art in Evaluation and Management. ISAKOS 2014. Alberto Gobbi, Joao Espregueira-Mendes, Norima Nakamura Editors
- [Background] Diederichs G, Issever AS, Scheffler S. MR imaging of patellar instability: injury patterns and assessment of risk factors. Radiographics. 2010 Jul-Aug;30(4):961-81. doi: 10.1148/rg.304095755. PMID 20631363
- [Background] Biedert RM. [Osteotomies]. Orthopade. 2008 Sep;37(9):872, 874-6, 878-80 passim. doi: 10.1007/s00132-008-1294-5. German. PMID 18682913
- [Background] Pache T, Meystre JL, Delgado-Martins H, Schnyder P. [Transplantation of the anterior tibial tubercle by the Elmslie-Trillat technic. Indications as a function of morphotype]. Rev Chir Orthop Reparatrice Appar Mot. 1985;71(6):359-64. French. PMID 4081137
- [Background] Rhee SJ, Pavlou G, Oakley J, Barlow D, Haddad F. Modern management of patellar instability. Int Orthop. 2012 Dec;36(12):2447-56. doi: 10.1007/s00264-012-1669-4. Epub 2012 Oct 7. PMID 23052278
- [Background] Guilbert S, Chassaing V, Radier C, Hulet C, Remy F, Chouteau J, Chotel F, Boisrenoult P, Sebilo A, Ferrua P, Ehkirch FP, Bertin D, Dejour D; French Arthroscopy Society (SFA). Axial MRI index of patellar engagement: a new method to assess patellar instability. Orthop Traumatol Surg Res. 2013 Dec;99(8 Suppl):S399-405. doi: 10.1016/j.otsr.2013.10.006. Epub 2013 Nov 20. PMID 24268843

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patellar Instability Group | Control Group Control
Started | 37 | 55
Completed | 37 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patellar Instability Group | Control Group Control | Total
Number analyzed (Participants) | 37 | 55 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 36 | 53 | 89
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years]
  mean | 28.6 (10.7) | 46 (14) | 39 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 14 | 36 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 37 | 55 | 92

OUTCOME MEASURES:

1. Primary Outcome: Existence of Tibial Tuberosity Torsion.
Description: This criteria will be considered relevant if it is associated with patellar dislocation. Existence Yes or No and measure of the torsion in degre on the IRM
Time Frame: 4 reviewers Assessment of 92 IRM of patients. Study data collection from April 2010 until december 2016. Patient duration follow up not applicable.
Population: Analysis based on the IRM available
Measure: Median (Inter-Quartile Range); unit: degre
Arm/Group | Patellar Instability Group | Control Group Control
Number analyzed (Participants) | 37 | 55
degre | 17.5 [13.0 to 23.9] | 5.3 [3.4 to 8.4]

2. Secondary Outcome: Measure of Patellar Tilt
Description: Patellar Tilt (yes or no), based on a patient IRM. Unit in degre.
Time Frame: 4 reviewers Assessment of 92 IRM of patients. Study data collection from April 2010 until december 2016. Patient duration follow up not applicable. Unit in degre
Population: Patients with IRM available.
Measure: Median (Inter-Quartile Range); unit: degre
Arm/Group | Patellar Instability Group | Control Group Control
Number analyzed (Participants) | 37 | 55
degre | 19.8 [13.8 to 27.6] | 5.3 [2.5 to 8.2]

3. Secondary Outcome: Distance TT-TG Tibial Tuberosity and Trochlear Groove
Description: distance between Tibial Tuberosity and Trochlear Groove
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: milimeters
Arm/Group | Patellar Instability Group | Control Group Control
Number analyzed (Participants) | 37 | 55
milimeters | 17 [12.2 to 20.1] | 8.4 [6.7 to 9.8]

ADVERSE EVENTS:
Time Frame: Not Applicable. Study consist in IRM reading. NO adverse events has been collected. Not applicable, retrospective study based on available IRM
Description: Not Applicable. Study consist in IRM reading. NO adverse events has been collected. Not applicable, retrospective study based on available IRM
Arm/Group | Patellar Instability Group | Control Group Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No